CLINICAL TRIAL: NCT04571515
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group, Dose-Response Study of MR-107A-01 in The Treatment of Post-Surgical Dental Pain
Brief Title: Dose-Response Study of MR-107A-01 in The Treatment of Post-Surgical Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MECC-TBZ-2001
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Pain; Postoperative Pain; Pain, Acute
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MR-107A-01 15 mg once in a 24-hour period (Experimental): Oral tablet one day of dosing
  Interventions: Drug: MR-107A-01
- MR-107A-01 10 mg once in a 24-hour period (Experimental): Oral tablet one day of dosing
  Interventions: Drug: MR-107A-01
- MR-107A-01 15 mg twice in a 24-hour period (Experimental): Oral tablet one day of dosing
  Interventions: Drug: MR-107A-01
- MR-107A-01 10 mg twice in a 24-hour period (Experimental): Oral tablet one day of dosing
  Interventions: Drug: MR-107A-01
- Placebo twice in a 24-hour period (Placebo Comparator): Placebo tablet one day of dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR-107A-01 — Oral tablet
  Arms: MR-107A-01 10 mg once in a 24-hour period; MR-107A-01 10 mg twice in a 24-hour period; MR-107A-01 15 mg once in a 24-hour period; MR-107A-01 15 mg twice in a 24-hour period
Drug: Placebo — Oral tablet
  Arms: Placebo twice in a 24-hour period

SUMMARY:
MR-107A-01 is being studied to investigate its efficacy, safety, and dose-response after dental surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Requirement for dental surgery for extraction of ≥2 x third molars, at least 1 of which involves partial or complete mandibular bony impaction.
3. Pain Intensity (PI) using a Numeric Pain Rating Scale (NPRS) ≥5 during the 5 hours following the end of surgery.
4. Rating of moderate or severe pain on a 4-point categorical pain rating scale (i.e., none, mild, moderate, severe) during the 5 hours following the end of surgery.

Exclusion Criteria:

1. Previously dosed with MR-107A-01.
2. Subject with known hypersensitivity to nonsteroidal antiinflammatory drugs (NSAIDs).
3. Active GI bleeding or a history of peptic ulcer disease, active inflammatory bowel disease, e.g., Crohn's Disease or ulcerative colitis, bleeding disorders that may affect coagulation.
4. Use of any investigational drug within 28 days, or 5 half-lives, prior to screening whichever is longer.
5. Use of medications with the potential to interact with MR-107A-01.
6. Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vogt, Study Director — MEDA Pharma GmbH & Co. KG (A Viatris Company)
Locations (1):
- Research Facility 101, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Started | 22 | 24 | 23 | 23 | 22
Completed | 21 | 24 | 23 | 23 | 19
Not Completed | 1 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — insufficient pain | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period | Total
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (2.17) | 19.2 (1.46) | 19.8 (2.37) | 19.4 (2.39) | 20.1 (2.41) | 19.7 (2.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 11 | 12 | 8 | 60
  Male | 10 | 6 | 12 | 11 | 13 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 6 | 7 | 3 | 23
  Not Hispanic or Latino | 19 | 19 | 17 | 16 | 18 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2 | 4
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 20 | 24 | 20 | 23 | 17 | 104
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Summed Pain Intensity Difference (SPID)
Description: Participants assessed Pain Intensity (PI) using a 0-10 numeric pain rating scale (NPRS) where 0 is no pain and 10 is worst pain imaginable. PI was assessed 17 times within 24 hours after the first study dose, and immediately before any rescue medication and/or at early termination. The participant's baseline PI was subtracted from the timepoint PI, to derive a Pain Intensity Difference (PID) for each timepoint. Overall Summed Pain Intensity Difference (SPID) measures pain intensity change relative to baseline over the 24 hour period after dosing, and corresponds to the Area Under the Curve (AUC) of the PID. In this study, higher positive Overall SPID indicates better pain improvement. Overall SPID could range from -120 to 240. Two hour windowed last observation carried forward was used as applicable where PI score obtained before a rescue medication replaced PI score for each timepoint within 2 hours following rescue dose.
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale * hours
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21
score on a scale * hours | 109.5 (32.82) | 111.8 (40.37) | 108.8 (33.85) | 108.6 (40.20) | 80.0 (39.78)
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.003, Emax; Mean Difference (Final Values) = 28.3, 95% CI 2-sided [9.9 to 46.6], Standard Error of Mean 9.25
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 29.6, 95% CI 2-sided [13.8 to 45.3], Standard Error of Mean 7.94
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 30.3, 95% CI 2-sided [14.4 to 46.2], Standard Error of Mean 8.04
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 31.1, 95% CI 2-sided [13.5 to 48.6], Standard Error of Mean 8.87

2. Secondary Outcome: Pain Intensity Using a Numeric Pain Rating Scale Utilizing 2-hour Windowed Last Observation Carried Forward (W2LOCF)
Description: 10 point scale, where 0 is no pain and 10 is the worst pain imaginable; 2-hour windowed last observation carried forward (W2LOCF) utilizes "pain right now" just prior to rescue medication use and censors subsequent pain intensity values for 2 hours when calculating SPIDs
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 22 | 21
score on a scale | 2.5 (1.86) | 2.1 (1.60) | 1.5 (1.34) | 2.3 (1.98) | 2.5 (2.39)
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.5 to 0.9], Standard Error of Mean 0.60
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.6], Standard Error of Mean 0.61
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.3], Standard Error of Mean 0.61

3. Secondary Outcome: Total Pain Relief
Description: Pain relief was assessed by participants using a 5 point scale, where 0 = none, 1 = slight, 2 = moderate, 3 = good or a lot, and 4 = complete. Pain relief was measured 17 times within 24 hours after the first study medication dose, and immediately before any rescue medication and/or at the time of early termination. Two-hour windowed last observation carried forward approach was used whereby the pain relief score obtained before a given rescue medication was carried forward to replace the pain relief scores collected at each observation timepoint within 2 hours following the rescue dose. Total pain relief (TOTPAR) had Areas Under the Curve (AUCs) calculated for each time point. The range for 24 hours post dose TOTPAR AUC was 0 to 96. Higher positive values indicate a better outcome with larger pain improvements.
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale * hours
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21
score on a scale * hours | 55.5 (12.31) | 57.3 (11.29) | 60.2 (13.48) | 56.6 (16.82) | 41.2 (17.05)
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 15.2, 95% CI 2-sided [7.3 to 23.1], Standard Error of Mean 3.99
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 16.1, 95% CI 2-sided [9.3 to 22.9], Standard Error of Mean 3.43
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 16.5, 95% CI 2-sided [9.7 to 23.4], Standard Error of Mean 3.47
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 17.1, 95% CI 2-sided [9.4 to 24.7], Standard Error of Mean 3.84

4. Secondary Outcome: Pain Relief: Number and Percentage of Subjects With Perceptible and Meaningful Pain Relief
Description: The time to onset of first perceptible relief was defined as the post dose time at which the subject first begins to feel pain relief. The time to meaningful pain relief was defined as the post dose time at which the subject begins to feel meaningful pain relief. The assessments of perceptible and meaningful pain relief were ceased when rescue medication was taken.
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21
Participants
  Perceptible Pain Relief | 15 | 22 | 16 | 19 | 10
  Meaningful Pain Relief | 10 | 17 | 13 | 15 | 3
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Perceptible Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.208, Log Rank
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Perceptible Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.005, Log Rank
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Perceptible Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.192, Log Rank
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Perceptible Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.067, Log Rank
Statistical Analysis 5: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Meaningful Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.059, Log Rank
Statistical Analysis 6: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Meaningful Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 7: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Meaningful Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.017, Log Rank
Statistical Analysis 8: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Time to Meaningful Pain Relief Subjects are censored at 24 hours if they do not report relief; Test type: Superiority; p = 0.002, Log Rank

5. Secondary Outcome: Patient's Global Assessment of Pain Control
Description: 5 point scale, where 0 is poor, 1 is fair, 2 is good, 3 is very good, and 4 is excellent Responder = 2 is good, 3 is very good, and 4 is excellent, Non-responder = 1 is fair, 0 is poor, and missing values
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21
Participants
  Responders | 14 | 16 | 18 | 13 | 7
  Non-responders | 7 | 8 | 5 | 10 | 14
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.051, Regression, Logistic
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.035, Regression, Logistic
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.016, Regression, Logistic
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.180, Regression, Logistic

6. Secondary Outcome: Rescue Medication Use
Description: Number of rescue medication doses
Time Frame: 24 hours after the first dose
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Medication doses
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
Number analyzed (Participants) | 21 | 24 | 23 | 23 | 21
Medication doses | 0.8 (1.03) | 0.8 (0.92) | 0.7 (0.70) | 0.7 (1.14) | 1.8 (1.58)
Statistical Analysis 1: Comparison: MR-107A-01 10 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.022, Wilcoxon Rank Sum
Statistical Analysis 2: Comparison: MR-107A-01 15 mg Once in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.028, Wilcoxon Rank Sum
Statistical Analysis 3: Comparison: MR-107A-01 10 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.007, Wilcoxon Rank Sum
Statistical Analysis 4: Comparison: MR-107A-01 15 mg Twice in a 24-hour Period vs Placebo Twice in a 24-hour Period; Test type: Superiority; p = 0.005, Wilcoxon Rank Sum

ADVERSE EVENTS:
Time Frame: Study period reporting of Adverse Events was up to 7 days post first dose. Subjects were reminded that AEs should be reported to the study staff up to 30 days after the last dose of study medication.
Description: An adverse event is any untoward medical occurrence in a patient/ clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment.
  An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory/ physical findings, symptom, or disease (new/ exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Arm/Group | MR-107A-01 10 mg Once in a 24-hour Period | MR-107A-01 15 mg Once in a 24-hour Period | MR-107A-01 10 mg Twice in a 24-hour Period | MR-107A-01 15 mg Twice in a 24-hour Period | Placebo Twice in a 24-hour Period
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24 | 0/23 | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 0/23 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 4/21 | 6/24 | 6/23 | 0/23 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MR-107A-01 10 mg Once in a 24-hour Period (N=21) | MR-107A-01 15 mg Once in a 24-hour Period (N=24) | MR-107A-01 10 mg Twice in a 24-hour Period (N=23) | MR-107A-01 15 mg Twice in a 24-hour Period (N=23) | Placebo Twice in a 24-hour Period (N=21)
Nausea (Gastrointestinal disorders) | 0 | 3 | 3 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT04571515/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT04571515/SAP_001.pdf